CLINICAL TRIAL: NCT05011734
Title: Rapid Postoperative Recovery (Fast-track) Pathway in Adolescent Idiopathic Scoliosis: a Pilot Study
Brief Title: Rapid Postoperative Recovery Pathway in Adolescent Idiopathic Scoliosis.
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: FAST-TRACK-IOR
Record Dates: First submitted 2021-07-28; First posted 2021-08-18 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Scoliosis Idiopathic
Keywords: Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fast Track recovery pathway — Multidisciplinary approach alongside the orthopedic surgeon

SUMMARY:
the study will evaluate the clinical outcomes of an intra- and postoperative fast-track protocol in patients undergoing instrumented posterior arthrodesis surgery for adolescent idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* Ages 14-18 years
* iagnosis of adolescent idiopathic scoliosis requiring an instrumented posterior arthrodesis surgical procedure
* Males and females.

Exclusion Criteria:

* spinal infection
* neoplastic diseases
* heart disease
* hypersensitivity to tranexamic acid
* history of coagulopathy and/or previous thromboembolic events
* severe renal failure

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents with idiopathic scoliosis treatable by surgical procedure
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Fast track protocol | at baseline (Day0)
  Evaluation of an intra- and post-operative fast-track protocol in terms of postoperative pain management.
Evaluation of the Fast track protocol | at baseline (Day0)
  Evaluation of an intra- and post-operative fast-track protocol in terms of duration/times of hospitalization
Evaluation of the Fast track protocol | at baseline (Day0)
  Evaluation of an intra- and post-operative fast-track protocol in terms of blood loss
Evaluation of the Fast track protocol | at baseline (Day0)
  Evaluation of an intra- and post-operative fast-track protocol in terms of patient education in early recovery of function.

SECONDARY OUTCOMES:
Surgical and clinical outcome | at baseline (Day0)
  evaluation of the hemocytometric examination (performed as per normal clinical practice).
Surgical and clinical outcome | at baseline (Day0)
  evaluation of the main circulating inflammatory mediators.
Surgical and clinical outcome | at baseline (Day0)
  evaluation of culture examinations on the surgical wound drainage fluid and microstructural analysis of the surgical drainage tube by scanning electron microscope.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Itituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang H, Tetteroo D, Arts JJC, Markopoulos P, Ito K. Quality of life of adolescent idiopathic scoliosis patients under brace treatment: a brief communication of literature review. Qual Life Res. 2021 Mar;30(3):703-711. doi: 10.1007/s11136-020-02671-7. Epub 2020 Oct 24. PMID 33098493
- [Result] Lee CS, Merchant S, Chidambaran V. Postoperative Pain Management in Pediatric Spinal Fusion Surgery for Idiopathic Scoliosis. Paediatr Drugs. 2020 Dec;22(6):575-601. doi: 10.1007/s40272-020-00423-1. Epub 2020 Oct 23. PMID 33094437
- [Result] Seki H, Ideno S, Ishihara T, Watanabe K, Matsumoto M, Morisaki H. Postoperative pain management in patients undergoing posterior spinal fusion for adolescent idiopathic scoliosis: a narrative review. Scoliosis Spinal Disord. 2018 Sep 12;13:17. doi: 10.1186/s13013-018-0165-z. eCollection 2018. PMID 30214945